CLINICAL TRIAL: NCT00619398
Title: A Multicenter, Randomized, Open Label, Parallel Study to Evaluate and Compare the Efficacy and Safety of FK506MR vs Prograf® in Stable Liver Transplantation Patients and a Pharmacokinetics Study
Brief Title: A Study to Evaluate and Compare the Efficacy and Safety of FK506MR vs Prograf® in Stable Liver Transplantation Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR4LTxCN02
Record Dates: First submitted 2008-01-23; First posted 2008-02-21 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Liver Transplantation
Keywords: FK506; tacrolimus; prograf; Liver transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Prograf
- 2 (Experimental)
  Interventions: Drug: FK506MR capsule

INTERVENTIONS:
Drug: Prograf — Oral
  Other Names: tacrolimus; FK506
  Arms: 1
Drug: FK506MR capsule — Oral
  Other Names: Advagraf; tacrolimus modified release capsule; MR4; Prograf XL
  Arms: 2

SUMMARY:
This study aims to evaluate and to compare the efficacy and safety of FK506MR with Prograf® in stable liver transplantation patients. It shall be demonstrated that FK506MR is non-inferior to Prograf® with regards to the efficacy and safety.

DETAILED DESCRIPTION:
A multicentre, randomized, open label, two parallel group study The patients will be randomized to MR4 group or Prograf® group. The treatment period is 3 months( 12 weeks).Patients randomized to MR4 group who complete 3 months treatment period will continue to use MR4 until MR4 commercial available or authority notification.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent with the date of the patient must be obtained
2. Patient is the recipient of a liver transplant from 6 to 24 months prior to enrollment
3. Patient is currently receiving Prograf or Prograf + MMF based immunosuppressive therapy
4. At screening the liver and kidney function of patient is stable (defined as Serum creatinine is normal and ALT or AST is <= 2 times the upper value of normal range)
5. Patient has the stable whole blood trough level concentration of Prograf (defined as tacrolimus trough concentrations of 2-10ng/ml measured 14 days prior to enrollment), and is clinically stable in the opinion of the investigator

Exclusion Criteria:

1. Patient has received an organ transplant other than a kidney
2. Patient has experienced any rejection episode within 90 days prior to enrollment in the study, any rejection episode within the last 6 months that required anti-lymphocyte antibody therapy
3. Patient is currently receiving other immunosuppressant therapy, eg. sirolimus
4. Patient with liver recurrent cancer, or metastasis, or other cancer
5. Patient has any unstable medical condition that could interfere with the study objectives
6. Patient is currently participating in another clinical trial and/or is taking or has been taking an investigational drug in the 30 days prior to enrollment
7. Patient is allergic macrolide antibiotics or tacrolimus
8. Patient has psychiatric disorder, in the opinion of the investigator, may invalidate communication with the investigator
9. Patient is currently receiving any medications, which is know to alter the CYP450 3A enzyme system (including grapefruit juice)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Event rate of patients with acute rejections | 12 Weeks

SECONDARY OUTCOMES:
Incidence of and time to acute rejections | 12 Weeks
Overall frequency of acute rejections | 12 Weeks
Rate of patients and graft survival following transplantation | 12 Weeks
Incidence of adverse events including laboratory assessments | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (6):
- China (6):
  - Beijing, Beijing Municipality
  - Guangzhou, Guangdong
  - Shenyang, Liaoning
  - Shanghai, Shanghai Municipality
  - Hangzhou, Zhejiang
  - Tianjing

IPD SHARING:
Plan to Share IPD: Undecided